CLINICAL TRIAL: NCT04296851
Title: The Chemopreventive Effect of Niclosamide in Patients With Familial Adenomatous Polyposis: Double Blinded Randomized Controlled Study
Brief Title: Niclosamide for Familial Adenomatous Polyposis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2017-0566
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Familial Adenomatous Polyposis
Keywords: chemoprevention; niclosamide; familial adenomatous polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Niclosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- niclosamide (Experimental): 650mg daily
  Interventions: Drug: Niclosamide
- placebo (Placebo Comparator): identical- appearing placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Niclosamide — The subjects will be randomly assigned in a 2:1 ratio to receive niclosamide or identical-appearing placebo tablets orally for 6 months: niclosamide 650mg once a day in arm 1, placebo once a day in arm 2.
  Arms: niclosamide
Drug: placebo — The subjects will be randomly assigned in a 2:1 ratio to receive niclosamide or identical-appearing placebo tablets orally for 6 months: niclosamide 650mg once a day in arm 1, placebo once a day in arm 2.
  Arms: placebo

SUMMARY:
Familial adenomatous polyposis (FAP) leads to adenomas and eventual adenocarcinomas in colon and less frequently, duodenum. Chemopreventive strategies have been studied in FAP patients to delay the development of adenomas and cancers. The non-steroidal anti-inflammatory drugs (NSAIDs) and selective cyclooxygenase-2 inhibitor have shown the regression of colorectal and duodenal adenomas in FAP patients. However, these drugs showed gastrointestinal damage and cardiovascular risks, and new preventive strategies are needed. Niclosamide, an anti-helminthic drug, has recently been suggested to have a suppressive effect on tumorigenesis via inhibition of Wnt pathway, and have no significant safety issues. The investigators devised a double-blind randomized controlled trial to evaluate the effect of niclosamide on polyps of colorectum and duodenum in FAP patients.

DETAILED DESCRIPTION:
This clinical trial is a double-blind randomized controlled trial to evaluate the effect of niclosamide on polyps of colorectum and duodenum in FAP patients. FAP patients, satisfied an enrollment criteria, will be randomly assigned in a 2:1 ratio to receive niclosamide (650 mg) or placebo tablets orally once a day for 6 months. The base-line and six-month endoscopic examination (colonoscopy/sigmoidoscopy and upper gastrointestinal endoscopy) will be recorded, and photographs will be taken at the tattoo-marked area. The number and size of polyps, and a qualitative assessment of the total extent of polyposis will be measured. If there is no significant improvement in any of the 12 initial cases (niclosamide 8: placebo 4), this trial will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Patients with familial adenomatous polyposis(FAP) who are 20 to 65 years of age.
* FAP patients who have colonic or duodenal polyp.
* FAP patients who have five or more polyps 2mm or more in diameter in endoscopic examination.

Exclusion Criteria:

* FAP patients who had a history of colectomy within the previous 12 months or need to undergo colectomy within 8 months after randomization.
* FAP patients with malignant disease, including colorectal cancer.
* FAP patients who used NSAIDs (non-steroidal anti-inflammatory drugs) or aspirin three or more times a week within 6 months of randomization.
* Pregnant or breast-feeding patients. 6. Patients with abnormal results of serum laboratory tests (renal function and liver function test).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Mean percentage change of the number and size of polyps in colon and/or duodenum. | After six-month administration of niclosamide/placebo
  At the base-line endoscopy (colonoscopy and upper gastrointestinal endoscopy), india-ink tattoo will be placed in the ascending colon, sigmoid colon/rectum, and duodenum. In case of the subjects with retained rectum after colectomy and ileorectal anastomosis, sigmoidoscopy will be performed. The base-line and six-month endoscopic examination will be recorded, and photographs will be taken at the tattoo-marked area and used for measurements of the number and size of polyps. The diameter of a polyp will be measured with the aid of biopsy forceps included in the photographic field, and only distinct polyps at least 2 mm in diameter will be counted.

SECONDARY OUTCOMES:
A qualitative assessment of the total extent of colorectal polyposis | After six-month administration of niclosamide/placebo
  A qualitative assessment of the total extent of colorectal polyposis will be conducted via video review(at base line and month 6) by two endoscopists experienced in the management of FAP, and scored as the same as, better than, or worse than base-line endoscopic findings, without the endoscopists' being aware of treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No